CLINICAL TRIAL: NCT00221000
Title: A Phase II, Multicenter, Randomized, Double-blind, "Sham" Pheresis-controlled, Study of Extracorporeal Photoimmune Therapy With UVADEX for the Treatment of Rheumatoid Arthritis in Patients Who Have an Inadequate Response to Disease Modifying Antirheumatic Drugs and Biological Agents
Brief Title: Safety and Efficacy of Extracorporeal Photoimmune Therapy With UVADEX for the Treatment of Rheumatoid Arthritis
Acronym: RA-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methoxsalen; Photopheresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methoxsalen
Procedure: Extracorporeal Photopheresis

SUMMARY:
Rheumatoid arthritis (RA) is a systemic autoimmune inflammatory disorder that can cause substantial pain and joint tenderness, significant joint damage, and serious disability. The treatment goals are minimization of the signs and symptoms of the disease, and the reduction of irreversible joint damage.

As the understanding of the pathophysiological mechanisms underlying RA is elucidated, the opportunity to target specific inflammatory processes with new therapies has improved. Rheumatoid arthritis is a T cell-mediated autoimmune disease and there are various therapies, including newer experimental therapies, which target either the activation of T cells or the neutralization of their effector mechanisms. These newer therapies have shown benefit in human and animal models of RA. Extracorporeal photoimmune therapy (ECP) has been shown to be safe and effective in the palliative treatment of the skin manifestations of cutaneous T cell lymphoma. Experimental studies have also demonstrated activity of ECP treatment in several T cell mediated diseases including graft versus-host disease, rejection after organ transplantation, and selected autoimmune diseases.

This study will evaluate a cell-based therapy (ECP) in patients who have an inadequate response to disease-modifying antirheumatic drugs (DMARDs) and biological agents to determine if ECP treatment can reduce the signs and symptoms of RA in this refractory patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of RA per the ACR criteria for the classification of RA.
* Patients must have moderately to severely active RA.

Moderately to severely active RA patients are defined as those patients meeting the following classification criteria, upon review by a physician, during screening: At least nine tender joints; At least six swollen joints;

PLUS (at least one of the following):

Morning stiffness, lasting greater than or equal to 45 minutes; Erythrocyte Sedimentation Rate greater than or equal to 28 mm/hour (ESR, to be evaluated at a local laboratory) or C reactive protein (CRP) greater than or equal to 15 mg/dL (to be evaluated at a central laboratory).

- Patients must have an inadequate response and continue to have moderately to severely active disease while on current or previous treatment with at least one agent from both of the following groups: methotrexate (greater than or equal to 15 mg/week, or maximum tolerated dose) or leflunomide (20 mg/day, or maximum tolerated dose) for at least 12 weeks prior to screening; etanercept ( greater than or equal to 25 mg/2 x week SC, or maximum tolerated dose) for at least 12 weeks prior to screening, infliximab (greater than or equal to 3 mg/kg IV, or maximum tolerated dose) for at least 14 weeks duration prior to screening, or adalimumab (greater than or equal to 40 mg SC every 2 weeks, or maximum tolerated dose) for at least 12 weeks prior to screening.

Note: In individual cases or in a country where access to anti TNF agents is limited or anti TNF agents are unavailable, the Investigator should document the reason for lack of availability of this treatment. Those patients who have not been treated with an anti-TNF agent would still be eligible for the study if they have failed treatment with at least two additional DMARDs, besides MTX and/or leflunomide. All patients may have also failed treatment with other biological agents or a protein A column.

* Patients who are not on oral corticosteroids. OR Patients who have been on a stable dose of oral corticosteroids at a prednisone equivalent dosage greater than or equal to 15 mg/day for at least 4 weeks prior to screening.
* Patients must have a platelet count greater than or equal to 100,000/cmm.
* Female patients must be one of the following: postmenopausal, surgically incapable of bearing children, practicing an acceptable method of birth control (acceptable methods may include hormonal contraceptives, intrauterine device, and spermicide and barrier). Abstinence or partner/spouse sterility may also qualify at the Investigator's discretion. If a female patient is of childbearing potential, she must have a negative urine pregnancy test at screening.
* Patients must be able and willing to comply with all study procedures.
* Patients must be willing to sign an ICF.
* Patients must be greater than or equal to 18 years of age.
* Patients must have a body weight greater than or equal to 40 kg (88 lb).

Exclusion Criteria:

* Patients who have a form of arthritis or arthropathy, other than RA, or any current inflammatory condition that might confound the assessments (e.g., other connective tissue diseases or Lyme disease).
* Patients who have been enrolled in any investigational therapy study for the treatment of RA within 4 weeks prior to the start of the Treatment Period, or patients who are scheduled to receive investigational therapies or a plasma based apheresis procedure (e.g., a protein A column) for the treatment of RA during the course of the study.
* Patients unable to tolerate the extracorporeal volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, severe chronic obstructive pulmonary disease, severe asthma, renal failure, or hepatic failure.
* Patients with a poor tolerability of venipuncture or a lack of adequate venous access for required treatments and blood sampling.

Note: Every attempt should be made to enroll patients who have adequate peripheral venous access.

* Patients who have a known hypersensitivity or allergy to psoralen (methoxsalen).
* Patients who have a known hypersensitivity or allergy to both heparin and citrate products.
* Patients who are taking any of the following permitted DMARDs and biological agents and have not been on a stable dose for the specific indicated periods of time prior to screening: MTX for at least 8 weeks; leflunomide for at least 8 weeks; infliximab for at least 14 weeks; etanercept for at least 12 weeks; adalimumab for at least 12 weeks.
* Patients who are taking any of the following permitted medications and have not been on a stable dose for at least 4 weeks prior to screening: NSAIDs; anakinra; hydroxychloroquine; chloroquine; sulfasalazine; D-penicillamine; gold salts; azathioprine; oral corticosteroids (greater than or equal to 15 mg/day, prednisone equivalent dose).
* Patients whom the Investigator believes cannot be maintained on stable doses of permitted concomitant RA medications throughout the Treatment Period.
* Patients who are taking any of the following prohibited medications: cyclophosphamide; chlorambucil; intramuscular (IM) or intravenous (IV) corticosteroid injection(s), within 4 weeks of screening; intra-articular corticosteroid injection(s) > 60 mg prednisone equivalent total dose, within 4 weeks of screening.
* Patients who have any known malignant disease (other than basal cell carcinoma) currently or within the last 5 years.
* Patients who have a pre-existing blood dyscrasia such as bone marrow hypoplasia, leukopenia, thrombocytopenia, significant anemia, or a coagulation disorder.
* Patients with a persistent or severe infection within 12 weeks of screening.
* Patients with a history of drug or alcohol abuse within 12 weeks of screening.
* Patients with impaired hepatic function at screening as shown by abnormal liver function tests (LFT; i.e., aspartate transaminase [AST] or alanine transaminase [ALT] levels > 2 x the upper limit of normal [ULN]).
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-08; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
ACR 20 | week 24 and week 28
  At least a 20% improvement of ACR 20 from baseline

SECONDARY OUTCOMES:
ACR 50 | week 24 and week 28
  Improvement of at least 50% from baseline on ACR 50

CONTACTS AND LOCATIONS:
Overall Officials: EDWARD KEYSTONE, MD, Principal Investigator — Rebecca MacDonald Centre for Arthritis
Locations (32):
- United States (10):
  - Carroll County Arthritis and Osteoporosis Center, Westminister, Maryland
  - Clinical Pharmacology Study Group, Worchester, Massachusetts
  - Morristown Memorial Hospital, Morristown, New Jersey
  - AAIR Research Center, Rochester, New York
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Rheumatology Associates, Providence, Rhode Island
  - UT Southwestern Medical Center, Dallas, Texas
  - Arthritis and Osteoporosis Center of South Texas, San Antonio, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- Royal Brisbane Hospital, Herston, Australia
- General Hospital of Vienna, Vienna, Austria
- Belgium (2):
  - Hospital Brugmann, Brussels
  - Limburgs Universitair Centrum, Diepenbeek
- Rebecca MacDonald Centre for Arthritis, Toronto, Ontario, Canada
- France (2):
  - CHRU de Lille, Lille
  - Hopital Edouard Herriot, Lyon
- Germany (7):
  - Franz von Prummer Klinik, Bad Brückenau
  - University of Charite Clinic for Rheumatology and Immunology, Berlin
  - Klinikum der Universitat zu Koln, Cologne
  - Medizinische Klinik III, Erlangen
  - Abt. Rheumatologie und Klinische Immunologie, Hamburg
  - Westfalische wilhelms-universitat Munster, Münster
  - Medizinische Klinik des Evangelischen Kranken, Oldenburg
- Italy (3):
  - Universita degli Studi di Firenze, Florence
  - Universita de Genova - Ospedale S. Martino, Genova
  - University of Siena-Italy, Siena
- OPD- Hospital Civil "Dr. Jaun I. Menchaca", Guadalajara, Jalisco, Mexico
- Reumatologicka ambulancia, Polinika, Bratislava, Slovakia
- South Africa (3):
  - South African National Blood Service, Bloemfontein
  - Christian Barnard Mermorial Hospital, Cape Town
  - D6 Rheumatology Clinic and E5 Hematology Unit, Cape Town